CLINICAL TRIAL: NCT02160678
Title: A Double-Blind,Randomized,Parallel-Group,Vehicle-Controlled,MulticenterStudy ComparingaGenericTazaroteneCream,0.1%toReference Listed Drug Tazorac® Cream, 0.1% and Both Active Treatments to Vehicle Control in the Treatment of Acne Vulgaris
Brief Title: Generic Tazarotene Cream, 0.1% in the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: G & W Laboratories Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SYM 2014-01
Record Dates: First submitted 2014-03-19; First posted 2014-06-11 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- Tazarotene Cream, 0.1 % (Active Comparator): Tazarotene Cream, 0.1 % (G & W Laboratories, Inc.) - test product
  Interventions: Drug: Tazarotene Cream, 0.1 %
- Tazorac Cream, 0.1% (Other): Tazorac Cream, 0.1% (Allergan, Inc.) - reference product
  Interventions: Drug: Tazorac Cream, 0.1%
- Vehicle (Placebo Comparator): Cream Vehicle (placebo) (G & W Laboratories, Inc.)- vehicle
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Vehicle — Cream Vehicle (placebo) (G & W Laboratories, Inc.)- vehicle
  Other Names: Placebo
  Arms: Vehicle
Drug: Tazarotene Cream, 0.1 % — Tazarotene Cream, 0.1 % (G & W Laboratories, Inc.) - test product
  Other Names: Active
  Arms: Tazarotene Cream, 0.1 %
Drug: Tazorac Cream, 0.1% — Tazorac Cream, 0.1% (Allergan, Inc.) - reference product
  Other Names: Reference Listed Drug
  Arms: Tazorac Cream, 0.1%

SUMMARY:
To compare the safety and efficacy profiles of Tazarotene Cream, 0.1 % to the reference listed drug Tazorac® (tazarotene) Cream, 0.1 % in order to demonstrate bioequivalence, and to demonstrate superiority of the 2 active creams over that of the cream vehicle (placebo) in the treatment of acne vulgaris.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, parallel-group, multicenter, double-blind study of Tazarotene Cream, 0.1% in subjects with acne vulgaris. Subjects will be assigned in a 1:1:1 ratio to test product, reference product, or cream vehicle. Subjects will be admitted into the study only after written informed consent has been obtained and all of the inclusion and none of the exclusion criteria have been met. Randomized subjects will apply the study medication once daily in the evening for 12 weeks (84 days).

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the study.
2. Be a healthy male or non-pregnant female aged ≥ 12 and ≤ 40 years of age, inclusive.
3. Have a clinical diagnosis of acne vulgaris, defined as having all of the following:

   1. On the face, ≥ 20 inflammatory lesions (papules and pustules)
   2. On the face, ≥ 25 non-inflammatory lesions (open and closed comedones)
   3. On the face, ≤ 2 nodulocystic lesions (nodules and cysts)
   4. Baseline IGA of acne severity grade 2, 3, or 4
4. Be in general good health and free from any clinically significant disease other than acne vulgaris that might interfere with the study evaluations.
5. Be willing to refrain from use of all other topical acne medications or antibiotics during the 12-week treatment period.
6. Be willing and able to understand and comply with the requirements of the study, apply the study medication as instructed, return for the required treatment period visits, comply with therapy prohibitions, and be able to complete the study.
7. Female subjects of childbearing potential (excluding women who are surgically sterilized or postmenopausal for at least 2 years) must have a negative urine pregnancy test (with a minimum sensitivity of at least 50 mIU/mL for human chorionic gonadotropin [hCG], begin treatment during a normal menstrual period and must agree to use a medically accepted method of contraception during the study. The following are considered acceptable methods of birth control for the purpose of this study: oral contraceptives, contraceptive patches, contraceptive implant, vaginal contraceptive, double barrier methods (e.g., condom and spermicide), contraceptive injection (Depo-Provera®), intrauterine device (IUD), hormonal IUD (Mirena®), and abstinence with a documented second acceptable method of birth control if the subject becomes sexually active. Subjects entering the study who are on hormonal contraceptives must have been on the method for at least 90 days prior to the study and continue the method for the duration of the study. Subjects who had used hormonal contraception and stopped must have stopped no less than 90 days prior to Visit 1/Day 1.
8. Be willing to limit sun exposure overall, maintain a reasonably constant exposure, and avoid use of tanning booths or other UV light sources during participation in the study.

Exclusion Criteria:

1. Females who are pregnant, breast feeding, planning a pregnancy, or who do not agree to use an acceptable form of birth control during the study.
2. Presence of any skin condition that would interfere with the diagnosis or assessment of acne vulgaris (e.g., on the face: rosacea, dermatitis, psoriasis, squamous cell carcinoma, eczema, acneiform eruptions caused by medications, steroid acne, steroid folliculitis, or bacterial folliculitis).
3. Currently has active cystic acne, acne conglobata, acne fulminans, secondary acne, or severe acne requiring more than topical treatment.
4. Currently has facial sunburn.
5. Received initial administrations of estrogens or oral contraceptives < 3 months (90 days) prior to baseline (Visit 1/Day 1), or discontinued estrogens or oral contraceptives < 3 months (90 days) prior to baseline. Use of such therapy must remain constant during the study.
6. Use of any treatment listing in Table 8.1 more recently than the indicated washout period prior to baseline (Visit 1/Day 1).
7. Need or intent to continue to use any treatment listed in Table 8.1 during the current study.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1741 (Actual)
Dates: Start 2014-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of equivalence of the test product to the reference product | Week 12
  The primary evaluation of equivalence will be through 2-sided 90% confidence intervals (CIs) about the ratio in mean percent reduction from baseline to Visit 4/Week 12 in the number of inflammatory and non-inflammatory lesions, respectively, of the test product to the reference product. These evaluations are based on a normal distribution adjusted for the effects of treatment group and site.
Evaluation of superiority | Week 12
  The primary evaluation of superiority will be conducted using an analysis of variance (ANOVA) model on the mean percent reduction in inflammatory and non-inflammatory lesions, respectively, with treatment and site as fixed effects. Contrasts will be performed to compare each active treatment with the vehicle cream.

SECONDARY OUTCOMES:
Proportion of subjects with a clinical response of "success" | Week 12
  The secondary efficacy endpoint will include the proportion of subjects with a clinical response of "success" at Visit 4/ Week 12. Success is defined as an Investigator's Global Assessment (IGA) score that is at least 2 grades less than the baseline assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bukhalo, MD, Principal Investigator — Altman Dermatology Associates
Locations (1):
- Altman Dermatology Associates, Arlington Hts., Illinois, United States